CLINICAL TRIAL: NCT06507059
Title: A Phase 3 Study Comparing Clinical Outcomes in People Living With HIV (PLHIV) With Suboptimal Adherence Treated With Injectable Long-acting Antiretrovirals Versus Oral Antiretrovirals
Brief Title: Outcomes of the PLHIV With Suboptimal Viral Suppression to Injectable Long-acting Antiretrovirals
Acronym: SUPLA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301496A3; MOHW113-CDC-C-114-000106 (Other Grant/Funding Number: Taiwan Centers for Disease Control)
Record Dates: First submitted 2024-07-07; First posted 2024-07-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection; Non-Adherence, Medication
Keywords: HIV-1, non-adherence
MeSH Terms: conditions — Medication Adherence | interventions — cabotegravir; Rilpivirine; cabotegravir, rilpivirine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Long-Acting Injectable Treatment Group (Experimental): Immediate switch to long-acting injectable antiretrovirals on enrollment
  Interventions: Drug: cabotegravir/rilpivirine (600mg/ 900mg)
- Delayed Long-Acting Injectable Treatment Group (Active Comparator): Keep on standard all-oral antiretrovirals on enrollment for 24 weeks, then switch to long-acting injectable antiretrovirals
  Interventions: Drug: Antiretroviral Combinations

INTERVENTIONS:
Drug: cabotegravir/rilpivirine (600mg/ 900mg) — Immediate switch from oral antiretroviral to long-acting injectables
  Other Names: Cabenuva
  Arms: Immediate Long-Acting Injectable Treatment Group
Drug: Antiretroviral Combinations — Standard all-oral antiretroviral combinations
  Arms: Delayed Long-Acting Injectable Treatment Group

SUMMARY:
This study aims to determine whether people living with HIV (PLHIV) with suboptimal medical adherence can achieve better viral suppression with long-acting antiretrovirals (LA) compared to all-oral antiretrovirals.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, active-controlled, superiority trial on 40 adult subjects who had been diagnosed to have HIV infection for at least 12 months before enrollment but with suboptimal viral suppression despite antiretroviral treatment (ART), with the latest HIV-1 viral load ≥ 200 copies/mL. Participants' eligibility will be assessed through a review of their medical records, and individuals with established resistance to cabotegravir or rilpivirine will be excluded. Enrolled participants will then be randomized 1:1 to either "Delayed Switch to LA Treatment Group" or "Immediate LA Treatment Group" on enrollment. The "Delayed Switch to LA Treatment Group" will also switch to LA on week 24. The proportion of participants with HIV-1 RNA <200 copies/mL at week 24 in the two study groups will be compared. Psychologic assessments including self-stigma and depression assessment will also be performed on day1, at week 24 and week 52.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the written informed consent form for male and female participants aged 18 and above.
* At the time of enrollment, diagnosed with HIV infection for a minimum of 12 months.
* Under oral antiretroviral treatment (ART), which can be irregular or interrupted, with the most recent viral load ≥ 200 copies/mL.
* Body weight ≥ 35Kg.
* Willing to maintain contact with the research team throughout the study (provide accurate and reachable phone numbers, social accounts like Line, or reliable contact information of family or friends).
* Willing to receive gluteal (buttocks) drug injections.
* Willing to transition back to oral medication or follow the recommended treatment prescription according to the then-current national treatment guidelines after discontinuation of long-acting injectable drugs.

Exclusion Criteria:

* For those currently undergoing oral antiretroviral therapy, who have started or restarted oral ART for less than six consecutive months before screening.
* Previously undergone HIV drug resistance testing and known to have resistance mutations to either cabotegravir or rilpivirine.
* Unable to commit to maintaining contact with the research team throughout the study.
* Individuals who cannot receive treatment for hepatitis B during the period of transitioning to long-acting injections, if they are hepatitis B carriers.
* Individuals with buttock fillers.
* Women who are planning to become pregnant, pregnant, or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV-1 RNA <200 copies/mL | Week 24
  Percentage of study participants with plasma HIV-1 RNA <200 copies/mL at week 24

SECONDARY OUTCOMES:
HIV-1 RNA <50 copies/mL | Week 24, week 52
  Percentage of study participants with plasma HIV-1 RNA <50 copies/mL at week 24, 52
HIV-1 RNA <200 copies/mL | Week 52
  Percentage of study participants with plasma HIV-1 RNA <200 copies/mL at week 52
Change of plasma HIV-1 viral load | Week 24, week 52
  Change of plasma HIV-1 RNA at week 24, 52
Change of CD4 count | Week 24, week 52
  Change of CD4 count at week 24, 52
Occurrence of HIV and non-HIV related conditions | Week 24, week 52
  Percentage of study participants with HIV and non-HIV related conditions occurrence
Lost F/U rate | up to week 96
  Lost follow-up rate at every target visit
Usage of outreach drug delivery service | up to week 52
  Percentage of study participants who use the outreach drug delivery service
Resistant variant emergence | Week 24, week 52
  Resistant variant emergence detection if HIV-1 viral load ≥200 copies/mL
Adverse events | Week 24, week 52
  Incidence and severity of adverse events (AEs)
Discontinuation due to AEs | Week 24, week 52
  Discontinuation due to AEs at week 24, 52
Change of depression score | Week 24, week 52
  Change of depression score at week 24, 52
Change of self-stigma score | Week 24, week 52
  Change of self-stigma score at week 24, 52
Change of metabolic parameters | Week 24, week 52
  Change of metabolic parameters (body weight, BMI) at week 24, 52

OTHER OUTCOMES:
Achieved ART trough level assessment | Week 52
  Use liquid chromatography- mass spectrometry to determine rilpivirine and cabotegravir concentrations in stored remaining plasma specimen collected at each visit
Change of acceptability score | Day1 (post-injection), week 24, 52 for the immediate LA treatment group; week 24 (post-injection), and week 52 for the delayed switch to LA group.
  Acceptability assessment for long-acting injectable antiretrovirals
Delayed injections | up to week 52
  Percentage of delayed injections (>7 days after the target visit)
HIV-1 RNA <50 copies/mL | Week 72, week 96
  Percentage of study participants with plasma HIV-1 RNA <50 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Nan-Yu Chen, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Chang Gung Memorial Hospital, Taipei, Taipei
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No